CLINICAL TRIAL: NCT00827996
Title: Open Label,Phase Two Study to Assess the Efficacy and Safety of Adalimumab in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: To Assess the Efficacy and Safety of Adalimumab in Subjects With Moderate to Severe Hidradenitis Suppurativa
Acronym: HIDRI2007
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida Academic Dermatology Centers (Other)
Collaborators: Abbott (Industry)
Responsible Party: Francisco A Kerdel,M.D, Florida Academic Dermatology Centers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIDRI2007
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Apocrine glands; abcesses
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: adalimumab — Subjects will be given subcutaneous injections at weeks 0 (160mg), 2 (80mg), and then every other week (40mg) until week 12

SUMMARY:
The trial is a 12-week phase 2 study. Subjects will be given subcutaneous injections at weeks 0 (160mg), 2 (80mg), and then every other week (40mg) until week 12 in subjects with moderate to severe hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

Subjects with moderate to severe HS as defined by a HSSI > 8 AND at least ONE of the following:

1. HS >1 year duration with multiple ER or doctors visits related to HS
2. Intralesional kenalog injection >5/year, however none within 2 weeks of entry
3. Failed systemic retinoids, but not within 3 months of entry
4. Failed at least one prior course of antibiotic therapy, which must not have been administered within 2 weeks of entry to the study (excluding the recommended antibiotic regimen given for evidence of active infection immediately before enrollment)
5. History of surgery (reconstructive), but not within 3 months of entry

Exclusion Criteria:

1. Women who are pregnant, nursing, or planning pregnancy within 6 months after the last injection (this includes father's who plan on fathering a child within 6 months after their last injection).
2. Use of other systemic anti-inflammatory medication except NSAIDs and low dose systemic steroids (equal or less than 10 mg daily prednisolone or equivalent).
3. If found to have an active infection, patients must have completed topical or oral antibiotic therapy at least 7 days before first injection.
4. Have a known history of serious infections (e.g., hepatitis, pneumonia or pyelonephritis) in the previous 3 months.
5. Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
6. Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (e.g., nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly.
7. Have a concomitant diagnosis or history of congestive heart failure.
8. Have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2008-08

PRIMARY OUTCOMES:
To assess the efficacy and safety of adalimumab in subjects with moderate to severe hidradenitis suppurativa. Efficacy will be evaluated using the included Hidradenitis Suppurativa Severity Index (HSSI). | 13 weeks

SECONDARY OUTCOMES:
To evaluate the role of TNF alpha in the pathogenesis of hidradenitis suppurativa. | 13 weeks
To evaluate the ability of adalimumab to maintain suppression of the disease. | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Kerdel, M.D, Principal Investigator — Florida Academic Dermatology Centers